CLINICAL TRIAL: NCT00485524
Title: A Retrospective Evaluation of the Utility of NIRS Compared With Serum Lactate Levels in Predicting Poor Post-Operative Outcome After Repair of Complex Congenital Heart Disease
Brief Title: Comparison of NIRS and Serum Lactate to Predict Poor Post-operative Outcomes
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 06-177
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2008-07

CONDITIONS: Congenital Disorders
Keywords: Near Infrared Spectroscopy; Serum Lactate Levels; post operative outcomes
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mortality after neonatal cardiac repair remains significant, and neonates who have undergone operative repair of congenital heart disease may experience sudden and unexpected demise. Most of these deaths occur within the first 72 hours and have been attributed to poor systemic cardiac output. The literature currently does not define an early and reliable predictor of poor post-operative outcome in children with congenital heart disease who have recently undergone surgery.

The investigator wishes to perform a retrospective chart review to independently define the predictive values of both NIRS score and serial serum lactate levels in the setting of early post-operative morbidity.

DETAILED DESCRIPTION:
The retrospective data will be collected on the NIRS score and serum levels within the first 72 hours, in the pediatric cardiac population that is less than one month of age requiring intra-operative cardiopulmonary bypass. This information will be reviewed from medical charts between January 1, 2002 and December 31, 2005 at Children's Healthcare of Atlanta, Egleston Hospital. We predict approximately 1000 charts will be reviewed.

The investigator wishes to evaluate the relationship of those levels with cardiac diagnosis, operation performed, post-operative course and outcome; poor outcome defined as initiation of ECMO or death.

The investigator then wishes to compare the predictive values of NIRS score and serial serum lactate levels in the above setting to assess their respective efficacies in post-operative cardiac intensive care. The investigator will collect the following information from the medical record:

Laboratory: NIRS Indices, serum pH, lactic acid, Co-ox, CBC, Chemistry) Diagnosis Surgical Procedure Incidence of re-operation Length of ICU Stay Length of Hospital Stay Complications Length of Ventilation (how many days on the ventilator) Medications Cross Clamp Time Bypass Time Echocardiogram data Cardiac Catheterization Data Vital Signs Monitored Hemodynamic Measures Final outcome (discharged versus ECMO or death)

Demographic data will be summarized for all subjects. For each patient summary statistics will include the mean, standard deviation, frequency distribution, minimum, maximum and range.

The investigator wishes to perform a retrospective chart review to independently define the predictive values of both NIRS score and serial serum lactate levels in the setting of early post-operative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Egleston Hospital, Children's Healthcare of Atlanta patients' charts
* Jan. 1, 2002 through Dec. 31,2005
* data collected on NIRS score and serum levels within the first 72 hours, in the pediatric cardiac population that is less than one month of age requiring intra-operative cardiopulmonary bypass.
* Exclusion Criteria:
* Those who do not meet inclusion criteria

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric cardiac population that is less than one month of age requiring intra-operative cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2002-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the relationship of serum lactate levels with cardiac diagnosis, operation performed, post-operative course and outcome. | within the first 72hr of intra-operative cardiopulmonary bypass

SECONDARY OUTCOMES:
Compare the predictive values of NIRS score and serum lactate levels in the above setting to assess their respective efficacies in post-operative cardiac intensive care. | within the first 72hr of intra-operative cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O Maher, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States